CLINICAL TRIAL: NCT05826288
Title: Design of a Patient-Centered Approach to Manage Bone Marrow Transplant Patients and CAR-T Cell Therapy in a Home Setting
Brief Title: Oncology Care at Home for BMT and CAR-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Reimagine Care (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-1832.cc
Record Dates: First submitted 2023-03-23; First posted 2023-04-24 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Leukemia
Keywords: Bone Marrow Transplant (BMT); Chimeric Antigen Receptor T-cell therapy (CAR-T)
MeSH Terms: conditions — Leukemia | interventions — Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post BMT or CAR-T patients receiving care at UCHealth (Experimental): Participants will be recruited for this study from among three discrete patient populations:
  * Allogeneic BMT patients receiving care at UCHealth who are planning to reside in the Denver metro area within 45 minutes of the Anschutz Medical Campus (AMC) for at least 90 days post-transplant.
  * Autologous BMT patients receiving care at UCHealth who are planning to reside in the Denver metro Area within 45 minutes of the AMC for at least 30 days post-transplant.
  * CAR-T patients receiving care at UCHealth who are planning to reside in the Denver metro area within 45 minutes of the AMC for at least 30 days post treatment.
  Interventions: Other: BioIntelliSense BioButton Rechargable; Other: Memora Health two-way patient engagement platform provided by RC

INTERVENTIONS:
Other: BioIntelliSense BioButton Rechargable — This study uses the BioIntelliSense BioButton Rechargeable for RPM, in combination with the BioSync mobile app on participants' mobile phones for data transmission, augmented by use of the BioHub as a backup transmission device. RPM monitoring of device data is accomplished through use of the AlertWatch software system.
  Other Names: Remote Patient Monitoring (RPM)
Other: Memora Health two-way patient engagement platform provided by RC — The Memora Health platform is designed to automate complex care workflows, making them simple for patients and clinicians to navigate. It utilizes a multi-modal communications system that primarily relies on two-way text messaging and artificial intelligence.

SUMMARY:
To assess the potential for successfully using technology-assisted in-home oncology care to provide improved care coordination and management, and appropriate referral to treatment for patients receiving bone marrow transplant (BMT) or chimeric antigen receptor (CAR) T-cell therapy (CAR-T). The technology-assisted in-home oncology care program includes remote patient monitoring (RPM), telemedicine, and home-based health care services.

DETAILED DESCRIPTION:
The objective of this study is to assess the potential for successfully using technology-assisted in-home oncology care to provide improved care coordination and management, and appropriate referral to treatment for patients receiving bone marrow transplant (BMT) or chimeric antigen receptor (CAR) T-cell therapy (CAR-T). The technology-assisted in-home oncology care program includes remote patient monitoring (RPM), telemedicine, and home-based health care services.

The study focuses on evaluating the technical feasibility, operational feasibility, and perceived patient, caregiver and healthcare provider experience of a combined package of technology-assisted in-home oncology care services to monitor for febrile neutropenia, infection, cyotokine release syndrome, neurotoxicity or other symptomatic episodes needing management up to 90 days post allogeneic BMT, up to 30 days post autologous BMT, and up to 30 days post CAR-T. It includes the following specific aims and hypotheses:

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years to 89 years old
* Bone marrow transplant recipients (allogeneic and autologous) or CAR-T patients
* Determined by care provider to be stable for discharge to home setting for outpatient care according to clinical practice standard operating procedures (SOPs)
* Residing in the Denver metro area for the duration of the study within 45 minutes of the AMC
* Has in-home caregiver support 24/7 (i.e., does not live alone)
* Has self-reported reliable telephone and home internet service and a stable wireless network
* Patient agrees to not submerge the BioButton Rechargeable device in more than 3 feet of water or submerge for longer than 30 minutes at a time.
* Patient owns or possesses, as the primary user with reliable daily access, a mobile device (iOS or Android) capable of running the study's mobile applications and accepting the terms and conditions
* Patient has SMS texting capacity and an unlimited texting plan or other plan sufficient for study text messaging without undue patient burden
* Patient is willing to complete and log a self-check of temperature twice daily and return the log to the study team at the end of the study
* Patient is willing to be available for the duration of the study
* Patient has access to reliable transportation to the hospital 24/7

Exclusion Criteria:

* Patients will be excluded from study participation if the PI or designated care provider believes study participation would not be in the patient's best interest for clinical reasons.
* Patients may also be excluded from study participation if in the opinion of the PI they have a medical condition that may impede their ability to adhere to the study protocol.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients reporting symptoms | 90 Days
  Determine the number of patients reporting symptoms via EPRO
Number of alerts generated through RPM systems | 30 days
Number of potential febrile events detected via RPM | 90 Days
Number of potential infections detected via RPM | 90 Days
Number of potential neurotoxicity events detected via RPM | 90 Days
Number of potential cytokine release syndrome (CRS) events detected via RPM | 90 Days
Number of febrile neutropenia events confirmed by clinical evaluation | 90 Days
Number of infections confirmed by clinical evaluation | 90 Days
Number of neurotoxicity events confirmed by clinical evaluation | 90 Days
Number of CRS events confirmed by clinical evaluation | 30 days
Number of tech support contacts received from patients/caregivers | 90 Days
Minutes RPM devices spent off-body | 90 Days

SECONDARY OUTCOMES:
Total number of patient interactions with RC | 90 Days
  Total patient interactions with RC, by type, including EPRO text message conversations, video visits, and phone calls
EPRO patient response rates | 90 Days
  The percentage of outbound text messages requesting a response that are responded to by persons activated on the program
Patient retention rate | 90 Days
  The percentage of patients that remain actively engaged with the program by exchanging at least one text message or having at least one telehealth encounter with the VCC per week
Number of calls escalated to CU/UCHealth for clinical evaluation and follow-up with study participants | 90 Days
Number of hospital admissions during study period | 90 Days
Length of stay for hospital admissions during study period | up to 90 days
Total days in hospital during study period | 90 Days
Number of emergency room visits during study period | 90 Days
Number of ICU admissions during study period | 90 Days

OTHER OUTCOMES:
Overall patient satisfaction | 90 days
  Number and percent of patients who report overall satisfaction with the intervention based on responses to survey items
Overall caregiver satisfaction | up to 90 days
  Number and percent of caregivers who report overall satisfaction with the intervention based on responses to survey items
Overall health care provider satisfaction | 90 days
  Number and percent of providers who report overall satisfaction with the intervention based on responses to survey items
Perceived quality of life | 90 days
  Number and percent of patients who report overall improvement in perceived quality of life in responses to survey items

CONTACTS AND LOCATIONS:
Overall Officials: Glen Peterson, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States